CLINICAL TRIAL: NCT06116084
Title: Randomized Controlled Study Evaluating the Efficacy of Hypnosis by Deportee Method Adapted to Nuclear Medicine
Brief Title: Randomized Controlled Study Evaluating the Efficacy of Hypnosis in Nuclear Medicine
Acronym: HYDEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Martine Louis, Prinicpal investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021PI059
Record Dates: First submitted 2022-01-21; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Myocarditis; Alzheimer Disease; Parkinson
MeSH Terms: conditions — Neoplasms; Myocarditis; Alzheimer Disease | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ericksonian hypnosis (Active Comparator): An Ericksonian hypnosis session given to patients during a scintigraphic or PET examination, in a conventional manner, i.e. the hypnotherapist (MERM) is close to the patient in the examination room at the time of the session and communicates with him/her without any special device dedicated to this purpose.
  Interventions: Other: Ericksonian Hypnosis
- Experimental hypnosis (Experimental): Hypnosis session with headphones and microphones
  Interventions: Other: Hypnosis

INTERVENTIONS:
Other: Ericksonian Hypnosis — An Ericksonian hypnosis session given to patients during a scintigraphic or PET examination, in a conventional manner, i.e. the hypnotherapist (MERM) is close to the patient in the examination room at the time of the session and communicates with him/her without any special device dedicated to this purpose.
  Arms: Ericksonian hypnosis
Other: Hypnosis — A hypnosis session given to patients during a scintigraphic or PET examination, in a remote manner, i.e. the hypnotherapist (MERM) is in the control room at the time of the session and communicates with the patient via a microphone and the patient has headphones.
  Arms: Experimental hypnosis

SUMMARY:
In Nuclear Medicine, the examinations are long (20-60 minutes) and the patients must remain immobile, sometimes fasting. The anxiety of the latter can lead to poor quality examinations and sometimes, although already injected with radioactive drugs, the patients refuse the examination. In imaging, the use of hypnosis (prior to the MRI examination or with the patient during a scintigraphic examination) is frequent due to the conformation of MRI or scintigraphic machines, particularly for claustrophobic patients (2-2.5% of cases).

Medical electroradiology manipulators (MERM) have been trained to practice Ericksonian hypnosis whose effectiveness in combating anxiety is no longer in question. Scientific studies by Faymonville et al, 2006 and Rainville et al, 2002, have shown the effectiveness of this method in managing anxiety using the simplified STAI-6 scale before and after hypnosis.

The dosimetric study of the MERM position would then be greatly modified in favor of a decrease in exposure targeted by the June 4, 2018 decree on personnel safety. The impact of whether or not the MERM is physically present near the patient would also be studied. If minimal, this will resolve the current contradiction between the quality of patient care delivered and the radiation protection imposed in nuclear medicine.

The investigators propose here a pilot study evaluating remote-delivered Ericksonian hypnosis versus conventionally-delivered Ericksonian hypnosis, which will allow for the sizing of a subsequent multicenter randomized non-inferiority controlled trial. Indeed, there is currently no data available on the non-inferiority margin of this technique.

DETAILED DESCRIPTION:
In Nuclear Medicine, the examinations are long (20-60 minutes) and the patients must remain immobile, sometimes fasting. The anxiety of the latter can lead to poor quality examinations and sometimes, although already injected with radioactive drugs, the patients refuse the examination. In imaging, the use of hypnosis (prior to the MRI examination or with the patient during a scintigraphic examination) is frequent due to the conformation of MRI or scintigraphic machines, particularly for claustrophobic patients (2-2.5% of cases).

Medical electroradiology manipulators (MERM) have been trained to practice Ericksonian hypnosis whose effectiveness in combating anxiety is no longer in question. Scientific studies by Faymonville and Rainville have shown the effectiveness of this method in managing anxiety using the simplified STAI-6 scale before and after hypnosis.

During nuclear medicine examinations, the proximity of MERMs to patients to practice conventional hypnosis results in significant exposure to radioactive radiation, which is not compatible with radiation protection guidelines. Some MERMs have been practicing hypnosis for several years, others are reluctant. However, exposure decreases as a function of the decrease in exposure time and the distance to the radioactive source. If the examination time cannot be modified, the distance to the patient could be by using an original method, remote hypnosis using a headset and microphone to provide Ericksonian hypnosis sessions in the same way as those provided in conventional sessions. The dosimetric study of the MERM position would then be greatly modified in favor of a decrease in exposure targeted by the June 4, 2018 decree on personnel safety. The impact of whether or not the MERM is physically present near the patient would also be studied. If minimal, this will resolve the current contradiction between the quality of patient care delivered and the radiation protection imposed in nuclear medicine.

The investigators propose here a pilot study evaluating remote-delivered Ericksonian hypnosis versus conventionally-delivered Ericksonian hypnosis, which will allow for the sizing of a subsequent multicenter randomized non-inferiority controlled trial. Indeed, there is currently no data available on the non-inferiority margin of this technique. This pilot study will also allow for extensive documentation of the implementation of the remote hypnosis technique and for any necessary adjustments to the intervention to ensure its feasibility, acceptability, and reproducibility in the subsequent trial.

The hypothesis is that the use of remote-assisted hypnosis in nuclear medicine reduces patient anxiety as much as conventional Ericksonian hypnosis, while limiting the radiation exposure of the MERMs.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for a scan or PET scan
* Patient with a score > 11 on the STAI-6 scale.
* Person, speaking and understanding French
* Having received complete information on the organization of the research and having signed the informed consent
* Age ≥ 18 years, and ≤ 80 years.
* Affiliated with a social security plan.

Exclusion Criteria:

* People who have taken an anxiolytic treatment before going to nuclear medicine.
* Persons referred for a neurological examination.
* People with cognitive or auditory problems, or with a major depressive episode.
* Persons with cardiac rhythm disorders (cardiac arrhythmias)
* Persons who cannot perform the examination for which they need a hypnosis session
* Women of childbearing age who do not have an effective means of contraception
* Person referred to in articles L. 1121-5, L. 1121-7 and L1121-8 of the public health code (pregnant woman, parturient or nursing mother, adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice, adult person unable to express his consent).
* Person deprived of liberty by a judicial or administrative decision, subject to psychiatric care under articles L. 3212-1 and L. 3213-1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Difference in anxiety score | 1 year
  Difference in anxiety score, measured using the STAI-6 score, of patients before and after scintigraphic or PET examination for each method of Ericksonian hypnosis.
  The scale is on 11. If the patient has a score lower than 11 he is not anxious, if the score is higher the patient is anxious.

SECONDARY OUTCOMES:
Clinical Efficacy of heart rate | 1 year
  Difference in heart rates (beats/min) of patients before and after scintigraphy or PET scan for each Ericksonian hypnosis method practiced by conventional method.
Clinical Efficacy of respiratory rate | 1 year
  Difference in respiratory rates (number of respiratory movements/min) of patients before and after scintigraphy or PET scan for each Ericksonian hypnosis method
Process evaluation of the intervention for the subsequent multicenter trial | 1 year
  Intervention dose
Process evaluation of the intervention for the subsequent multicenter trial | 1 year
  Fidelity of the intervention to the protocol (by semi-directed interview conducted by a psychologist researcher with the manipulators to explore the hypnotherapist's experience of the session, and by quality criteria for the completion of the hypnosis session) ;
Process evaluation of the intervention for the subsequent multicenter trial | 1 year
  Target attainment (user satisfaction at the end of the examination, and by semi-structured interview conducted by a psychologist researcher to explore the patient's experience of the hypnosis session); adaptation (during semi-structured interviews with the manipulators).
Impact mechanisms | 1 year
  safety (manipulators operational dosimetry readings before and after each hypnosis session (µSv/h)), manipulators satisfaction at the end of each examination, quality criteria for performing the scan.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Louis, Principal Investigator — m.louis2@chru-nancy.fr
Locations (1):
- Nancy Hospital, Vandœuvre-lès-Nancy, France